CLINICAL TRIAL: NCT00534755
Title: Prospective & Retrospective Data Collection of Breast Cancer Cases From 2000 to Present
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RAC#2051-029
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Breast database (Other): Database
  Interventions: Other: Breast Cancer database

INTERVENTIONS:
Other: Breast Cancer database — prospective breast cancer database

SUMMARY:
Prospective & Retrospective data collection of breast cancer cases from 2000 to present

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2005-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Database | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Dahish Ajarim, MD, Principal Investigator — KFSH&RC
Locations (1):
- KFSH&RC, Riyadh, Saudi Arabia